CLINICAL TRIAL: NCT02344199
Title: A Non-interventional, Multicenter, Observational Clinical Trial to Assess Eplerenone Treatment in Patients With Heart Failure.
Brief Title: Eplerenone in Heart Failure Treatment
Acronym: INOSET
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-PLR-EL-55
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure; Acute Myocardial Infarction; Hypertension
MeSH Terms: conditions — Heart Failure; Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Beta-blockers should be administered to all patients with heart failure stage II to IV according to NYHA.Beta-blockers reduce mortality and hospitalizations and improve the operational phase for all categories of patients with heart failure. Since beta-blockers, only carvedilol, metoprolol, bisoprolol and recently nevimpololi have shown these benefits and so, only they have evidence to be provided.

Eplerenone is indicated, in addition to conventional therapy, for reducing the risk of cardiovascular mortality and morbidity in stable patients with left ventricular dysfunction (LVEF ≤ 40%) and clinically proven heart failure after recent myocardial infarction.

DETAILED DESCRIPTION:
Heart Failure (HF) As heart failure is defined as a complex clinical syndrome that can result from any structural or functional cardiac disorder and affects the ability of the ventricle to accept or eject blood. Its incidence is increasing in recent years in the Western world. It is estimated that 6% - 10% of the population over 65 suffers from heart failure. The clinical picture of heart failure is shortness of breath, fatigue tolerance restriction and fluid retention that can lead to pulmonary congestion or peripheral edema. These symptoms and signs are not required to appear all at once in each patient. Some patients simply have a reduced exercise tolerance, while others dominate the swelling and do not report dyspnea or fatigue. For the diagnosis of heart failure is necessary apart from the existence of symptoms objective confirmation cardiac dysfunction, preferably by echocardiography, or more specialized and less available methods, such as magnetic resonance imaging heart and radionuclide ventriculography.

Coronary heart disease is nowadays the dominant cause of heart failure, as 65-70% of patients with heart failure suffer from coronary disease. The cardiomyopathies and especially dilated, is the cause of heart failure in 20% of cases. The myocarditis, hyperthyroidism and abuse of ethanol, are responsible for a significant number of patients with type distending heart failure. Hypertension and valvular dominated in the past, occupy small percentage today as heart failure causes. The heart failure can be divided into right or left, depending on whether the predominant symptoms resulting from congestion of systemic or pulmonary veins, respectively. Moreover, heart failure is separated into systolic or diastolic depending on whether systolic or diastolic performance of the left ventricle is affected. In most patients with systolic heart failure and diastolic dysfunction coexist. However, in 30% of patients with heart failure is pure diastolic dysfunction.

For the diagnosis of heart failure with diastolic dysfunction criteria require:

1. In the presence of signs and symptoms of heart failure
2. ejection fraction of the left ventricle> 45%
3. the presence of one of three types of abnormal left ventricular filling during diastole (relaxation extension, restrictive type).

There are four operating stages depending on the symptoms of patients with heart failure, according to the classification in NYHA (New York Heart Association). At the operational stage I patients have symptoms of heart failure at a high level of exercise, beyond the ordinary. In stage II, the symptoms appear in a regular exercise level at stage III in small fatigue, while in stage IV symptoms occur at rest, so that patients are unable to look after themselves. Medication and diet can alter the operating phase which is the patient, without any significant change occurs in ventricular performance. It is particularly interesting that there is little correlation between symptoms and systolic left ventricular performance as expressed by the ejection fraction. Thus, patients with low ejection fraction <25% can be virtually asymptomatic, while others slightly influenced ejection fraction have serious discomfort. Changes of abdominal diatasimotitas of pericardial voltage, any valvular deficiencies and especially the function of the right ventricle are those factors which together with systolic left ventricular performance determine the occurrence or not of the symptoms of heart failure patients. In heart failure the function of the left ventricle is gradually worsening even in the absence of new effect damaging agent. This is the famous remodeling (Cardiac Remodeling) of the left ventricle, during which the investigators dilatation, hypertrophy and more spherical the shape. Thus, the mechanical performance of the ventricle decreases, increasing the mitral insufficiency due to distension of the mitral annulus, and increases the parietal stress. Ventricular remodeling contribute to continuous deterioration of symptoms, despite any treatment. The activation of the neurohormonal system proved to be the most important factor in why the cardiac remodeling and the unfavorable development of heart failure. Patients with heart failure have in their plasma levels of noradrenaline, angiotensin II, aldosterone, endothelin and cytokines which may act deleteriously on the structure and functioning of the heart. The mobilization of neurohormonal mechanisms in heart failure causes fluid retention and sodium, peripheral vasoconstriction, myocardial fibrosis and toxic effect on myocardial cells, creating a vicious cycle of deteriorating architecture and performance of the failing heart.

Ejection Fraction

The relation between stroke volume, which is extruded from the left ventricle and the starting end diastole filling volume gives a measure of the contractile function of the left ventricle. Each patient with known cardiovascular disease should be subject to assessment of left ventricular function by measuring ejection fraction. Several studies have demonstrated that when the ejection fraction (LVEF), which measures the ability of the heart to eject blood into the aorta, not exceed 40% (natural rate ^ 50%) increased dramatically postinfarction mortality. The ejection fraction is a reliable prognostic indicator can be calculated by ultrasonography. The reduced ejection fraction is associated with an increased risk of life-threatening arrhythmias, heart failure and death. A low ejection fraction, particularly after myocardial infarction, is a strong indication for the administration of beta-blockers, as many studies have shown that administration of these drugs significantly reduces cardiovascular mortality.

Rationale of the study

This study intends to recruit within 6 months of clinical practice in the Greek reality regarding the data administration of eplerenone in addition to standard therapy including beta-blockers, to reduce the risk of cardiovascular mortality and morbidity in stable patients with dysfunction left ventricle (LVEF ≤ 40%) and clinically proven heart failure after recent myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Eligible ages for the study:> 18 years
* Patients who are to receive eprelenone according to standard clinical practice
* Patients with heart failure of ischemic / non-ischemic etiology
* Patients receiving standard therapy including beta-blockers, to reduce the risk of cardiovascular mortality and morbidity
* Stable patients
* Patients with left ventricular dysfunction (LVEF ≤ 40%)
* Patients with clinically proven heart failure after recent myocardial infarction.
* Patients who have fully understood the study protocol and signed the consent form

Exclusion Criteria:

* Patients <18 years
* Hypersensitivity to eplerenone in any of the excipients
* Patients with a serum potassium level> 5,0 mmol / L at the start of therapy
* Patients with moderate to severe renal impairment (creatinine clearance <50 mL / min)
* Patients with severe hepatic impairment (Child-Pugh class C)
* Patients taking diuretics guard potassium loss or strong inhibitors of CYP3A4 (eg itraconazole, ketoconazole, ritonavir, nelfinavir, clarithromycin, telithromycin and nefazodone)
* Patients who have not fully understood the study protocol and have not signed the consent form

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Heart Failure
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Levels of Potassium (K) | 6 months

SECONDARY OUTCOMES:
Safety assessed by number of Adverse Events reported | 6 months
Potassium Levels (K) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Parissis, MD, Principal Investigator — Cardiology Department, Attikon University Hospital of Athens
Locations (3):
- Greece (3):
  - Cardiology University Clinic, Alexandroupoli, Alexandroupolis
  - Gennimatas General State Hospital, Athens, Attica
  - 2nd Cardiology Department,, University of Athens, Attikon Hospital, Haidari, Athens

REFERENCES:
- [Background] Preiss D, van Veldhuisen DJ, Sattar N, Krum H, Swedberg K, Shi H, Vincent J, Pocock SJ, Pitt B, Zannad F, McMurray JJ. Eplerenone and new-onset diabetes in patients with mild heart failure: results from the Eplerenone in Mild Patients Hospitalization and Survival Study in Heart Failure (EMPHASIS-HF). Eur J Heart Fail. 2012 Aug;14(8):909-15. doi: 10.1093/eurjhf/hfs067. Epub 2012 May 19. PMID 22611047
- [Background] Ademi Z, Pasupathi K, Krum H, Liew D. Cost effectiveness of eplerenone in patients with chronic heart failure. Am J Cardiovasc Drugs. 2014 Jun;14(3):209-16. doi: 10.1007/s40256-014-0066-3. PMID 24610254
- [Background] Rossignol P, Dobre D, McMurray JJ, Swedberg K, Krum H, van Veldhuisen DJ, Shi H, Messig M, Vincent J, Girerd N, Bakris G, Pitt B, Zannad F. Incidence, determinants, and prognostic significance of hyperkalemia and worsening renal function in patients with heart failure receiving the mineralocorticoid receptor antagonist eplerenone or placebo in addition to optimal medical therapy: results from the Eplerenone in Mild Patients Hospitalization and Survival Study in Heart Failure (EMPHASIS-HF). Circ Heart Fail. 2014 Jan;7(1):51-8. doi: 10.1161/CIRCHEARTFAILURE.113.000792. Epub 2013 Dec 2. PMID 24297687
- [Background] Collier TJ, Pocock SJ, McMurray JJ, Zannad F, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pitt B. The impact of eplerenone at different levels of risk in patients with systolic heart failure and mild symptoms: insight from a novel risk score for prognosis derived from the EMPHASIS-HF trial. Eur Heart J. 2013 Sep;34(36):2823-9. doi: 10.1093/eurheartj/eht247. Epub 2013 Jul 17. PMID 23864130
- [Background] Eschalier R, McMurray JJ, Swedberg K, van Veldhuisen DJ, Krum H, Pocock SJ, Shi H, Vincent J, Rossignol P, Zannad F, Pitt B; EMPHASIS-HF Investigators. Safety and efficacy of eplerenone in patients at high risk for hyperkalemia and/or worsening renal function: analyses of the EMPHASIS-HF study subgroups (Eplerenone in Mild Patients Hospitalization And SurvIval Study in Heart Failure). J Am Coll Cardiol. 2013 Oct 22;62(17):1585-93. doi: 10.1016/j.jacc.2013.04.086. Epub 2013 Jun 27. PMID 23810881
- [Background] Rogers JK, McMurray JJ, Pocock SJ, Zannad F, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pitt B. Eplerenone in patients with systolic heart failure and mild symptoms: analysis of repeat hospitalizations. Circulation. 2012 Nov 6;126(19):2317-23. doi: 10.1161/CIRCULATIONAHA.112.110536. Epub 2012 Oct 5. PMID 23042980
- [Background] Rywik TM. [Summary of the article: Zannad F, McMurray JJV, Krum H et al.; for the EMPHASIS-HF Study Group. Eplerenone in patients with systolic heart failure and mild symptoms. N Engl J Med, 2011; 364: 11-21]. Kardiol Pol. 2011;69(6):631-2. No abstract available. Polish. PMID 21678313
- [Background] Zannad F, McMurray JJ, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pocock SJ, Pitt B; EMPHASIS-HF Study Group. Eplerenone in patients with systolic heart failure and mild symptoms. N Engl J Med. 2011 Jan 6;364(1):11-21. doi: 10.1056/NEJMoa1009492. Epub 2010 Nov 14. PMID 21073363